CLINICAL TRIAL: NCT02366234
Title: Symptomatic Treatment of Distal Tubercle Fractures of the Scaphoid
Status: Withdrawn | Type: Observational
Why Stopped: The investigator left the institution so the study was terminated.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Haaglanden Medical Centre (Other); Skane University Hospital (Other); Ghaem Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Chief of Hand and Upper Extremity Service, Massachusetts General Hospital
Other Study IDs: 2014P002670
Record Dates: First submitted 2015-02-06; First posted 2015-02-19 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Distal Tubercle Fractures of the Scaphoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fracture of Distal Tubercle of Scaphoid: Questionnaires
  * Quick DASH after trauma (< 2 weeks)
  * 11-point ordinal measure of overall pain intensity 6 months after trauma
  * 11-point ordinal measure of satisfaction with treatment 6 months after trauma

SUMMARY:
AIM:

The aim of this study is to assess whether patients with an acute distal tubercle fracture of the scaphoid treated with a removable brace for 4 to 6 weeks have the same level of symptoms and disability 6 months after injury as the average for the normal population.

NULL HYPOTHESIS:

Patients with an acute distal tubercle fracture of the scaphoid have Quick DASH (Disabilities of the Arm Shoulder and Hand) scores at or above the population norm (a score of 13 in Norway and 10.9 in the United States) 6 months after injury when treated symptomatically with a removable brace.

DETAILED DESCRIPTION:
Fractures of the distal scaphoid tubercle are uncommon and seem relatively benign. Not a lot is known in literature about this specific type of avulsion fracture and the treatment. Some surgeons recommend a cast for 4 to 6 weeks while others treat their patients with a removable brace. The only non-union reported in literature is Jonssen who published a case in 1990 about a non-union of a tubercle fracture in a patient with repeated trauma. Kraus et al studied 81 cases of acute scaphoid fractures and found 4 cases of tubercle avulsion fractures in this group. We suspect some patients will not seek care for this condition as it hurts for a bit and then causes no problems.

Response variables:

* Quick DASH measured 6 months after injury
* 11-point ordinal measure of overall pain intensity 6 months after trauma

Explanatory variables:

* Socio-demographics
* Age, sex, ethnicity, race, marital status, education, work status
* Questionnaires
* Quick DASH after trauma (< 2 weeks)
* 11-point ordinal measure of overall pain intensity 6 months after trauma
* 11-point ordinal measure of satisfaction with treatment 6 months after trauma

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Fracture of the distal tubercle of the scaphoid on radiographs
* Interval between injury and diagnosis of less than 2 months
* English or Spanish fluency and literacy

Exclusion Criteria:

* Pregnant women
* Inability to complete enrollment forms due to any mental status or language problems (e.g. dementia, head injury, overall illness)
* Patients with other fractures or injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with distal tubercle fracture of the scaphoid
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Disability with use of QuickDASH | 2 weeks

SECONDARY OUTCOMES:
Overall Pain Intensity | 6 months
  Pain Intensity measured with an 11-point ordinal measure of overall pain intensity 6 months after trauma
Satisfaction with Treatment | 6 months
  Satisfaction measured with an 11-point ordinal measure of satisfaction with treatment 6 months after trauma

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD PhD, Principal Investigator — Massachusetts General Hospital